CLINICAL TRIAL: NCT06157190
Title: Incorporating Wearable Technology for Enhanced Rehabilitation Monitoring After Hip and Knee Replacement
Acronym: MOVEUP-WT
Status: Completed | Type: Observational
Sponsor: PXL University College (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Other Study IDs: PXLuc
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis; Osteoarthritis, Hip
Keywords: wearable technology; rehabilitation monitoring
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with knee replacement: The knee replacement patient cohort in this study consists of individuals who underwent Total Knee Arthroplasty (TKA) and utilized the moveUP digital application for at least six weeks post-surgery. The criteria include:
  Total Knee Arthroplasty (TKA): Individuals who had surgical intervention for total knee replacement.
  moveUP Digital Application Usage: Patients actively engaged with the moveUP digital therapies platform, using the associated application for rehabilitation. The application aids and monitors the recovery process.
  Post-Surgery Duration of Six Weeks: To be part of the study, patients in this cohort used the digital application for a minimum of six weeks after knee replacement surgery. This duration aims to evaluate the effectiveness of technology-assisted rehabilitation during the critical early recovery phase.
  Interventions: Other: Unsupervised monitoring
- patients with hip replacement: The hip replacement cohort likely comprises individuals who had total hip arthroplasty. Similar to the knee replacement cohort, inclusion criteria may involve using the moveUP digital application for at least six post-surgery weeks. Characteristics include:
  Total Hip Arthroplasty (THA): Patients underwent surgical intervention for total hip replacement.
  moveUP Digital Application Usage: Cohort members actively engaged with the moveUP digital therapies platform, utilizing the associated app for post-surgery rehabilitation.
  Post-Surgery Duration of Six Weeks: To join the study, patients likely used the digital application for a minimum of six weeks post-hip replacement surgery. This period helps assess technology-assisted rehabilitation effectiveness during early recovery.
  Interventions: Other: Unsupervised monitoring

INTERVENTIONS:
Other: Unsupervised monitoring — This study introduces technology-assisted rehabilitation for patients post-total hip or knee arthroplasty, utilizing wearable sensors and mobile health tech. The intervention includes:
  Technology-Assisted Rehabilitation: Utilizing wearable sensors and mobile health technologies, the intervention promotes unsupervised, real-world assessments after total hip or knee replacement. It shifts from traditional supervised clinical assessments. The moveUP digital therapies platform, featuring a dedicated mobile app, acts as the primary interface for patients in rehabilitation.
  Digital Biomarkers: The intervention involves gathering digital biomarkers from wearable sensors and mobile health tech. These biomarkers offer continuous, objective measurements of patients' biological and physiological data. Examples include mobility and activity level data.

SUMMARY:
This study focuses on the impact of osteoarthritis (OA), a leading cause of disability among older adults, with the hip and knee joints being particularly affected. The rise in OA prevalence is attributed to factors such as aging and increasing obesity rates. Post-surgery rehabilitation, especially after total hip or knee replacement, traditionally relies on supervised clinical assessments, which have limitations in capturing real-world experiences. The study aims to explore the integration of technology-assisted rehabilitation, utilizing wearable sensors and mobile health technologies, for unsupervised, real-world assessments. The use of digital biomarkers collected from these technologies offers continuous, objective measurements of patients' biological and physiological data. The research employs a dataset from moveUP digital therapies, including patients who underwent total knee arthroplasty, utilizing a digital application for at least six weeks post-surgery.

Key objectives include evaluating the potential of automated unsupervised assessments in providing a holistic understanding of patient progression during rehabilitation. The study utilizes mixed models for statistical analysis, examining outcomes such as steps per day, 6-minute walk test, and peak 1 minute. Results indicate differences in recovery trajectories between hip and knee patients, with variations based on gender and type of prosthesis.

DETAILED DESCRIPTION:
Data Source:

This retrospective observational study utilized anonymized and depersonalized data from the moveUP digital therapies database (moveUP solution, Brussels, Belgium). The database encompasses information from patients who underwent hip and knee arthroplasty across Belgium, France, and the Netherlands. A cohort of 1144 patients who underwent elective total knee arthroplasty was selected based on their use of the digital application for a minimum of 6 weeks post-surgery, with completion of preoperative patient-reported outcome measures. Written informed consent for the scientific use of anonymized data was obtained from each patient. Regulatory guidelines were adhered to, and no institutional review board (IRB) approval was required, given the use of anonymized patient-level data.

Recording Device and Outcomes:

All data collection occurred through the moveUP® application, a registered medical device operating on a smart virtual platform designed for digital monitoring. This platform comprises a patient-facing mobile application and a web-based dashboard utilized by care providers. Objective data, including the number of steps per day and steps per minute, were collected using a commercial activity tracker (Garmin Vivofit 4) worn 24/7 by patients throughout the rehabilitation period. Patient-reported outcomes, such as the Oxford Knee Score, Forgotten Joint Score (FJS), Hip Osteoarthritis Outcome score (KOOS), Knee Osteoarthritis Outcome score (KOOS), UCLA Activity Scale (UCLA), and the EuroQol 5-Dimension (EQ5D), were measured before surgery and at various intervals up to two years post-surgery through the app.

Statistical Analysis:

We analyzed outcomes using mixed models for both knee and hip patients, treating values from each day as repeated measures. The model incorporated fixed effects related to recovery, days after surgery, age, gender, and the interaction between recovery and days. Our analysis employed fixed effects for recovery, days after surgery, and their interaction, with baseline measures normalized for comparability. Time needed to differentiate between recovery statuses was computed along with associated 95% confidence intervals. Statistical analyses were conducted at a significance level of 0.05 using RStudio (version 2023.09.0) with R version 4.4.2 and the LME4 package for mixed effect models.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Hip or Knee Replacement surgery
* minimum 18 years of age
* Patient has emailadres
* use of application for at least 6 weeks postop
* completion of preoperative questionnaire

Exclusion Criteria:

* Patient younger than 18 years of age
* no emailadres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with Osteoarthritis (OA): The study focuses on individuals affected by osteoarthritis, a common degenerative joint condition.
  * Age Group:
  * Underwent Hip or Knee Replacement Surgery: The population includes individuals who have undergone either total hip arthroplasty or total knee arthroplasty.
  * Geographical Distribution: The dataset used for the study is from moveUP digital therapies and includes patients from Belgium, France, and the Netherlands. Therefore, the study population is likely diverse, representing patients from these regions.
  * Technology-Engaged Individuals:The study population engaged with technology-assisted rehabilitation through the moveUP digital therapies platform.
  * Minimum Post-Surgery Duration: Patients engaged with the technology-assisted rehabilitation for a minimum of six weeks post-surgery, indicating a focus on the early stages of the recovery process.
Sampling Method: Non-Probability Sample
Enrollment: 1144 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
steps per day | pre and 6 weeks post surgery
  This parameter represents the daily step count of patients. Monitoring steps per day is a common metric for assessing mobility and physical activity during rehabilitation.
6 minute walking test | pre and 6 weeks post surgery
  he 6-minute walk test is a standard measure of functional capacity and endurance. Patients are assessed on the distance they can walk in six minutes, providing valuable information about their cardiovascular and musculoskeletal function
Peak 1 Minute | pre and 6 weeks post surgery
  Refers to the walking performance measured during a one-minute interval
Intensity | pre and 6 weeks post surgery
  intensity of physical activity, specifically focusing on activities classified as moderate-to-vigorous. This parameter provides information about the intensity of patients' physical efforts during rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Move Up, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided